CLINICAL TRIAL: NCT01020279
Title: Multiple-dose, Randomized, Subject and Observer Blinded, Placebo-controlled, Double-dummy Study of Epicutaneously Applied Ketoprofen Transfersome® Gel With or Without Combination With Oral Celecoxib for the Treatment of Muscle Pain Induced by Eccentric Exercise
Brief Title: Study of Epicutaneously Applied Ketoprofen Transfersome® Gel With or Without Combination With Oral Celecoxib for the Treatment of Muscle Pain Induced by Eccentric Exercise
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: X-pert Med GmbH (Industry)
Responsible Party: Dipl. med. Ilka Rother, X-pert Med GmbH
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: XPM-023
Record Dates: First submitted 2009-11-09; First posted 2009-11-25 (Estimated); Last update posted 2010-06-28 (Estimated); Status verified 2010-06

CONDITIONS: Musculoskeletal Pain
Keywords: muscle pain; model
MeSH Terms: conditions — Musculoskeletal Pain; Myalgia | interventions — Celecoxib; Ketoprofen

STUDY DESIGN:
Who Masked: Participant

ARMS (2):
- Parallel Group A (Other): Celecoxib 200 mg (Active Comparator) ; Ketoprofen in Transfersome® Gel (Experimental); Placebo Gel (Placebo Drug)
  Interventions: Drug: Celecoxib, Ketoprofen
- Parallel Group B (Other): oral Placebo (Placebo Comparator); Ketoprofen in Transfersome® Gel (Experimental); Placebo Gel (Placebo Drug)
  Interventions: Drug: Ketoprofen

INTERVENTIONS:
Drug: Celecoxib, Ketoprofen — Ketoprofen in Transfersome® gel, 2 g gel on the calf, 4 g gel on the quadriceps, b.i.d.
  Celecoxib, 200 mg, one capsule b.i.d.
  Arms: Parallel Group A
Drug: Ketoprofen — Placebo gel, 2 g gel on the calf, 4 g gel on the quadriceps, b.i.d. Oral placebo, one capsule b.i.d
  Arms: Parallel Group B

SUMMARY:
1. Comparison of the effect of ketoprofen Transfersome® gel (KTG) to placebo gel (PG) on muscle pain of the calf caused by eccentric contractions
2. Comparison of the effect of KTG to celecoxib (CE) on muscle pain of the calf caused by eccentric contractions
3. Comparison of the effect of celecoxib (CE) to oral placebo (OP) on muscle pain of the calf caused by eccentric contractions

ELIGIBILITY:
Inclusion Criteria:

* Signed and dated informed consent prior to participation
* Subjects in good health as determined by the Investigator
* Age 18-55
* Willing to abstain from any physical therapy, hard physical work, exercise or sauna during the study observation period (Screening to Final Visit)
* For females, subjects of childbearing potential (including peri-menopausal women who have had a menstrual period within 1 year) must be using appropriate birth control (defined as a method which results in a low failure rate, i.e., less than 1% per year when used consistently and correctly, such as implants, injectables, some intrauterine contraceptive devices (IUDs), sexual abstinence, or a vasectomized partner). Oral contraceptive medications are allowed in this study. Female subjects, who are surgically sterile (bilateral tubal ligation, bilateral oophorectomy or hysterectomy) are also allowed for participation

Exclusion Criteria:

* Participation in another clinical study within the last 30 days and during the study
* Subjects who are inmates of psychiatric wards, prisons, or other state institutions
* Investigator or any other team member involved directly or indirectly in the conduct of the clinical study
* Pregnancy or lactation
* Alcohol or drug abuse
* Malignancy within the past 2 years with the exception of in situ removal of basal cell carcinoma
* Skin lesions, dermatological diseases or tattoo in the treatment areas
* Known hypersensitivity or allergy (including photoallergy) to NSAID´s including celecoxib, sulfonamides and ingredients used in pharmaceutical products and cosmetics including galactose
* Varicosis, thrombophlebitis and other vascular disorders of the lower extremities
* Major traumatic lesions (e.g. fracture, tendon or muscle ruptures) of the musculo-skeletal system of the lower limbs
* Pain conditions which might interfere with pain rating during the study, e.g. neuropathic pain
* Significant neurological or psychiatric symptoms resulting in disorientation, memory impairment, or inability to report accurately (e.g. Alzheimer's disease or schizophrenia or other psychosis), that in the investigator's opinion may affect efficacy or safety assessments or may compromise subject safety during the study
* Systemic lupus erythematodes, mixed connective tissue disease
* Major heart disease / uncontrollable hypertension
* Peripheral arterial disease and/or cerebrovascular disease
* History of stroke or myocardial infarction
* GFR < 30 ml/min
* ALT and/or AST levels ≥ 5 times the ULN
* Chronic obstructive pulmonary disease including asthma bronchiale
* Coagulopathy or bleeding diathesis, or concomitant use of anticoagulants including low dose aspirin
* History of pancreatitis or peptic ulcers
* Inflammatory GI disease (e.g. M. Crohn, colitis ulcerosa)
* Reflux esophagitis requiring treatment
* Any other analgesic therapy including cough and cold drugs containing analgesic properties as well as any other substance used for the treatment of pain during the study observation period (Screening to final Visit)
* Any other drug that might alter pain perception like CNS active drugs

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 82 (Actual)
Dates: Start 2009-10; Study Completion 2010-01 (Actual)

PRIMARY OUTCOMES:
Pain during muscle contraction | Day 7

SECONDARY OUTCOMES:
Pain during rest | Day 7
Surface temperature | Day 7
Volume of the lower leg | Day 7

CONTACTS AND LOCATIONS:
Locations (1):
- X-pert Med GmbH, Jena, Germany